CLINICAL TRIAL: NCT06050759
Title: C-Reactive Protein / Albumin Ratio as a Predictive Inflammatory Marker for Postoperative Systemic Inflammatory Response Syndrome and/or Sepsis in Polytraumatized Patients in ICU
Brief Title: CRP/Albumin Ratio as a Predictive Inflammatory Marker for Postoperative SIRS and/or Sepsis
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ahmed Samir Said Salem, Assistant Lecturer of Anaesthesia and Intensive care, Ain Shams University
Other Study IDs: MD134/2023
Record Dates: First submitted 2023-09-16; First posted 2023-09-22 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Crp
Keywords: CRP/ALBUMIN Ratio; Systemic inflammatory response syndrome; Sepsis; postoperative
MeSH Terms: conditions — Systemic Inflammatory Response Syndrome; Sepsis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: CRP and Albumin level in blood sample — CRP and Albumin levels will be measured from blood samples of the patients to determine CRP/Albumin Ratio

SUMMARY:
The goal of this observational study is to determine the value of CRP/Albumin Ratio as an inflammatory marker for predicting the development of postoperative Systemic Inflammatory Response Syndrome and/or Sepsis in polytraumatized patients admitted to Intensive care unit.

The main question it aims to answer is whether CRP/Albumin Ratio can be used as predictive inflammatory marker for postoperative Systemic Inflammatory Response Syndrome and/or Sepsis or not.

DETAILED DESCRIPTION:
The development of postoperative Systemic Inflammatory Response Syndrome (SIRS) or Sepsis is a very serious complication that has been associated with high morbidity, mortality, and increased length of inpatient stay.

Sepsis is a life-threatening organ dysfunction caused by a dysregulated host response to infection.

As surgical interventions lead to well-understood metabolic, neuroendocrine, and immune responses, the stress responses to surgery contribute to increased postoperative complications mostly caused by increased levels of Pro-inflammatory cytokines in response to surgical injury, which leads to changes of circulating acute phase proteins, such as albumin and C-reactive protein (CRP).

The CRP to albumin ratio (CAR) is a new index calculated by dividing CRP by the albumin level. It has been assumed to have predictive value in determining morbidity and mortality in many critical diseases.

ELIGIBILITY:
Inclusion Criteria:

* Patients classified by American Society of Anesthesiologists physical status (ASA) as I to III.
* Both sex.
* Aged ≥ 18 years old.
* Polytraumatized patients (fulfilling the 'New Berlin definition' of Polytrauma patient which includes Abbreviated Injury Scale (AIS) ≥3 for two or more different body regions with one or more of the following five physiological variables: Disturbed level of consciousness, hypotension, coagulopathy, acidosis and age >70y).
* Admitted to Intensive Care Unit preoperatively or postoperatively. • Surgical intervention within 48 hours of the onset of Trauma.

Exclusion Criteria:

* Patients who used immunosuppressive therapy and chemotherapy.
* Patients with known hematological disorders or malignancy.
* Patients with known liver cirrhosis classified as Child- Pugh C ( serum Albumin < 2.8 mg/dl or International Normalized Ratio > 2.2 ) (Tsoris , et al.,2023) or liver cell failure.
* Patients receiving Albumin Supplementation during the period of the study.
* Age < 18y.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Patients classified by American Society of Anesthesiologists physical status (ASA) as I to III.
  * Both sex.
  * Aged ≥ 18 years old.
  * Polytraumatized patients (fulfilling the 'New Berlin definition' of Polytrauma patient which includes Abbreviated Injury Scale (AIS) ≥3 for two or more different body regions with one or more of the following five physiological variables: Disturbed level of consciousness, hypotension, coagulopathy, acidosis and age >70y).
  * Admitted to Intensive Care Unit preoperatively or postoperatively. • Surgical intervention within 48 hours of the onset of Trauma.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Evaluate the relation of CRP/ albumin ratio to the prediction of postoperative SIRS or sepsis in polytrauma patients. | The patients will be evaluated for 5 days postoperatively
  Evaluate the relation of CRP/ albumin ratio to the prediction of postoperative SIRS or sepsis in polytrauma patients.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Samir, Doctor, Principal Investigator — Faculty of Medicine Ain shams University
Locations (1):
- AinShams University Specialized Hospital, Cairo, Abbasia, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rhodes A, Evans LE, Alhazzani W, Levy MM, Antonelli M, Ferrer R, Kumar A, Sevransky JE, Sprung CL, Nunnally ME, Rochwerg B, Rubenfeld GD, Angus DC, Annane D, Beale RJ, Bellinghan GJ, Bernard GR, Chiche JD, Coopersmith C, De Backer DP, French CJ, Fujishima S, Gerlach H, Hidalgo JL, Hollenberg SM, Jones AE, Karnad DR, Kleinpell RM, Koh Y, Lisboa TC, Machado FR, Marini JJ, Marshall JC, Mazuski JE, McIntyre LA, McLean AS, Mehta S, Moreno RP, Myburgh J, Navalesi P, Nishida O, Osborn TM, Perner A, Plunkett CM, Ranieri M, Schorr CA, Seckel MA, Seymour CW, Shieh L, Shukri KA, Simpson SQ, Singer M, Thompson BT, Townsend SR, Van der Poll T, Vincent JL, Wiersinga WJ, Zimmerman JL, Dellinger RP. Surviving Sepsis Campaign: International Guidelines for Management of Sepsis and Septic Shock: 2016. Intensive Care Med. 2017 Mar;43(3):304-377. doi: 10.1007/s00134-017-4683-6. Epub 2017 Jan 18. PMID 28101605
- [Background] Ge X, Cao Y, Wang H, Ding C, Tian H, Zhang X, Gong J, Zhu W, Li N. Diagnostic accuracy of the postoperative ratio of C-reactive protein to albumin for complications after colorectal surgery. World J Surg Oncol. 2017 Jan 10;15(1):15. doi: 10.1186/s12957-016-1092-1. PMID 28069031
- [Background] Iyengar KP, Venkatesan AS, Jain VK, Shashidhara MK, Elbana H, Botchu R. Risks in the Management of Polytrauma Patients: Clinical Insights. Orthop Res Rev. 2023 Mar 21;15:27-38. doi: 10.2147/ORR.S340532. eCollection 2023. PMID 36974036
- [Background] Kim MH, Ahn JY, Song JE, Choi H, Ann HW, Kim JK, Kim JH, Jeon YD, Kim SB, Jeong SJ, Ku NS, Han SH, Song YG, Choi JY, Kim YS, Kim JM. The C-Reactive Protein/Albumin Ratio as an Independent Predictor of Mortality in Patients with Severe Sepsis or Septic Shock Treated with Early Goal-Directed Therapy. PLoS One. 2015 Jul 9;10(7):e0132109. doi: 10.1371/journal.pone.0132109. eCollection 2015. PMID 26158725
- [Background] Singh B, Goyal A, Patel BC. C-Reactive Protein: Clinical Relevance and Interpretation. 2025 May 3. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK441843/ PMID 28722873
- [Background] Pape HC, Moore EE, McKinley T, Sauaia A. Pathophysiology in patients with polytrauma. Injury. 2022 Jul;53(7):2400-2412. doi: 10.1016/j.injury.2022.04.009. Epub 2022 May 14. PMID 35577600
- [Background] Proctor MJ, Horgan PG, Talwar D, Fletcher CD, Morrison DS, McMillan DC. Optimization of the systemic inflammation-based Glasgow prognostic score: a Glasgow Inflammation Outcome Study. Cancer. 2013 Jun 15;119(12):2325-32. doi: 10.1002/cncr.28018. Epub 2013 Apr 10. PMID 23575969
- [Background] Tsoris A, Marlar CA. Use Of The Child Pugh Score In Liver Disease. 2023 Mar 13. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK542308/ PMID 31194448
- [Background] Uzum Y, Turkkan E. Predictivity of CRP, Albumin, and CRP to Albumin Ratio on the Development of Intensive Care Requirement, Mortality, and Disease Severity in COVID-19. Cureus. 2023 Jan 10;15(1):e33600. doi: 10.7759/cureus.33600. eCollection 2023 Jan. PMID 36788868